CLINICAL TRIAL: NCT02636751
Title: Effects of a Tele-prehabilitation Program or an In-person Prehabilitation Program Compared to a Usual Care Control Group in Participants Awaiting Total Hip or Knee Arthroplasty: A Pilot Single Blind Randomized Controlled Trial
Brief Title: Effects of Tele- or In-person Prehabilitation in Candidates Awaiting Total Hip or Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Montréal (Other)
Collaborators: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, François Desmeules, Professor, School of Rehabilitation, University of Montreal, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DOIP2015
Record Dates: First submitted 2015-12-14; First posted 2015-12-22 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Osteoarthritis
Keywords: Prehabilitation; Telemedicine; Osteoarthritis; Arthroplasty; Hip; Knee
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- In-person prehabilitation group (Experimental): The participants in this group will receive a 12-week rehabilitation program (2x/week) including, education, stretching, strengthening, proprioceptive exercises of the lower limb and cardiovascular training using low-impact activities, in addition to walking aid adjustment. General information about pain control, such as ice application and medication usage will also be provided
  Interventions: Behavioral: 12-week prehabilitation program; Device: Walking aid adjustment; Behavioral: Information about pain control
- Tele-prehabilitation group (Experimental): The participants in this group will receive a 12-week rehabilitation program (2x/week) including, education, stretching, strengthening, proprioceptive exercises of the lower limb and cardiovascular training using low-impact activities, in addition to walking aid adjustment using a telecommunication software (Reacts®, Facetime® or Skype®). General information about pain control, such as ice application and medication usage will also be provided.
  Interventions: Behavioral: 12-week prehabilitation program; Device: Walking aid adjustment; Behavioral: Information about pain control
- Usual care group (Active Comparator): The participants in this group will be provided with the hospital's usual documentation before total joint arthroplasties, consisting of information regarding the pre- and post-surgery course and medication.
  Interventions: Device: Walking aid adjustment; Behavioral: Information about pain control

INTERVENTIONS:
Behavioral: 12-week prehabilitation program — stretching, strengthening, proprioceptive exercises of the lower limb and cardiovascular training using low-impact activities
  Arms: In-person prehabilitation group; Tele-prehabilitation group
Device: Walking aid adjustment — Walking aid adjustment
Behavioral: Information about pain control — General information about pain control, such as ice application and medication usage

SUMMARY:
This pilot single blind randomized controlled trial aims therefore to evaluate the feasibility and the impact on pain and disabilities of a telerehabilitation prehabilitation program for patients awaiting a total joint (hip or knee) arthroplasty compared to in-person prehabilitation or to usual care.

DETAILED DESCRIPTION:
BACKGROUND

Osteoarthritis (OA) is a very common disorder that affects almost every Canadian over 65 years of age. Future estimations indicate the incidence of OA will increase by at least 26% over the next 30 years in Canada. Hip and knee are the most affected joints by OA and these conditions incur important disability. Lower limb OA is initially treated conservatively with therapeutic interventions such as physical activity modification, exercise, weight control, and medication. Surgical interventions such as total joint arthroplasty (TJA) have been proven a treatment of choice for the most severe cases. However, the accessibility to such surgery often comes up against long wait lists, and prolonged wait time may lead to deleterious effects on the health status and quality of life of the awaiting patients.

Prehabilitation refers to education and exercising before a surgery. Attention to prehabilitation has increased in the last decade and a growing body of evidence suggests that it could have a positive effect on postoperative outcomes and may reduce disabilities before and after surgery for a number of conditions. In the context of prehabilitation for TJA, trials have already shown that a rehabilitation exercise program before a TJA could lead to a shorter hospitalisation length of stay, in addition to increased muscle strength and range of motion following a total hip or knee arthroplasty. However, results concerning the longer-term effects of prehabilitation after a TJA tend to be inconsistent and further research is actually needed to better understand the effects of prehabilitation over the post-surgical course.

As the aging population and the constant increase in chronic diseases keep pressuring the healthcare systems worldwide, lack of resources tends to lengthen wait time for surgery like TJA. Long wait times for such medical interventions have a negative impact on pain, function and quality of life. Policymakers have therefore been searching for a care optimisation strategy to improve healthcare accessibility to prehabilitation.

Among the solutions stands the use of technology to help deliver more efficiently rehabilitation services or to improve access to these types of care. Telerehabilitation has gained increased recognition and it is defined as the provision of rehabilitation services at a distance, using information and communication technologies. Previous studies have already shown that telerehabilitation programs are feasible in a home-care setting.

Tousignant et al. demonstrated that a telerehabilitation program was as efficient and less expensive than conventional physiotherapy after a total knee arthroplasty (TKA). Bedra et al. qualified as viable a home-based telerehabilitation program after a hip fracture, while Anton et al. demonstrated that a Kinect™-based system can be an adjuvant to physiotherapy after a total hip replacement.

Those programs present good opportunities for optimising the delivery of care in community rehabilitation, especially by increasing the number of patients seen in a single day, by reducing medical costs and travel time, and by providing access to medical care otherwise unavailable in rural areas. However, no study, to our knowledge, analysed the outcome of telerehabilitation before proceeding to a total joint replacement.

This pilot single blind randomized controlled trial aims therefore to evaluate the feasibility and the impact on pain and disabilities of a telerehabilitation prehabilitation program for patients awaiting a total joint (hip or knee) arthroplasty compared to in-person prehabilitation or to usual care. Our hypothesis is that a 12-week prehabilitation program will significantly increase functional mobility and quality of life for the subjects in the experimental groups, but not in the control group.

EXAMINATION PROCEDURE AND RANDOMIZATION

During the baseline evaluation at the Maisonneuve-Rosemont Research Center, eligible participants will complete a questionnaire covering sociodemographic status, comorbidities, and medication usage. Patients will be asked to fill in four French validated self-reported questionnaires: the Lower Extremity Functional Scale (LEFS-CF), the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC-CF), the Short Form Health Survey (SF-36-CF) and a Global Rating of Change Scale (GRC-CF). Three physical functional performance measures will also be collected: the self-paced walk (SPW), the timed up-and-go (TUG) and timed stair tests (ST). These tests are oriented toward activities of daily living and have been validated with a geriatric population. They are reliable, reproducible, and responsive to change. They also have widely been used for measuring the outcomes of patients undergoing a TJA. An online version of the questionnaires using the Survey Monkey® platform or a paper version will be provided to the participants. Finally, a logbook will be given to the participants. They will be asked to record the exercises executed at home, including the number of series and repetitions, in addition to the medication intake. This logbook will allow a monitoring of the compliance rate to the programs and also the advent of any adverse effects.

Patients will then be randomly assigned to the control group or to one of the two experimental groups. An independent research assistant, blind to the baseline evaluation results, will open the randomization envelope indicating the participant's assignment to a group. A random number generator will be used to establish randomization lists prior to the initiation of the study. A member of the research team, not involved with data collection, will generate the randomization list. Blocked randomization of 6 will be used to make sure that three equal groups of 12 subjects participants are obtained.

Participants will be reassessed at 12 weeks by a blind research assistant, after the completion of the interventions. The same evaluation tools as at baseline will be used, according to a standardized procedure. A satisfaction questionnaire about the telecommunication software experience will be filled by participants and therapists who used a telecommunication software.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years;
2. Waiting for a TKA or a THA
3. Suffering from severe OA of hip or knee
4. Quebec resident covered by the Régie de l'assurance maladie du Québec (Quebec public healthcare insurance)
5. Speaks French
6. Has a high-speed internet connection.

Exclusion Criteria:

1. Suffering from inflammatory arthritis
2. Scheduled for a bilateral surgery
3. Has had a lower limb surgery in the past 6 months
4. Scheduled for a revision of a previous TKA or THA
5. Planned for a wide acetabular head hip prosthesis or a hip articular resurfacing
6. Receiving a compensation from Quebec Commission de la santé et de la sécurité du travail (government insurer for workers and employers)
7. Suffering from a severe psychiatric neurologic or cardiac disorder, or other types of disorders that could interfere with the rehabilitation program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-10 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change in Lower Extremity Functional Scale (LEFS) | At Baseline and 12 weeks after baseline
  20-item questionnaire. Each item is rated on a five-point scale (0= extreme difficulty or unable to perform activity, 4= no difficulty); total scores range from 0 to 80, and lower scores represent greater difficulty.

SECONDARY OUTCOMES:
Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) | At Baseline and 12 weeks after baseline
  Self-administered questionnaire. 24 items divided into 3 subscales: pain (5 items), stiffness (2 items) and physical function (17 items). Each item is scored on a five-point scale according to difficulty experienced (0 = none and 4 = extremely difficult(40).
Change in Short Form (36) Health Survey | At Baseline and 12 weeks after baseline
  self-administered generic health status measure questionnaire. It calculates 8 multi-item scales (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health) and 2 summary scales, the physical component summary (PCS) and the mental component summary (MCS).
Change in Global Rating of Change scale (GRC) | At Baseline and 12 weeks after baseline
  designed to quantify a patient's perceived improvement or deterioration over time. Using an 11-point GRC scale, ranging from -5 (a great deal worse) to 0 (about the same) to +5 (a great deal better), participants will be asked to answer the following question: "Overall, has there been any change in your condition since the initial evaluation done at the beginning of your rehabilitation program? Please indicate if there has been any change in your condition by choosing one of the following options".
Change in Timed Up and Go (TUG) | At Baseline and 12 weeks after baseline
  test that assesses mobility, balance, walking ability, and fall risk in older adults. The patient sits in a chair with his/her back against the chair back. On the command "go", the patient rises from the chair, walks 3 meters at a comfortable and safe pace, turns, walks back to the chair and sits down. Timing begins at the instruction "go" and stops when the patient is seated. Time in seconds is the outcome of the test.
Change in StairTest (ST) | At Baseline and 12 weeks after baseline
  Patients are asked to ascend and descend 8 stairs (step height 18.5 cm) in their usual manner, at a safe and comfortable pace. Use of a gait aide and/or of the handrail is allowed as needed(30). Time in seconds is the outcome of the test.
Change in Self-Paced Walk test | At Baseline and 12 weeks after baseline
  Patients are required to walk two lengths of a 20 m indoor course in response to the instructions ''walk as quickly as you can without overexerting yourself.'' Usual gait aides are allowed as needed.
Satisfaction questionnaire | At 12 weeks after baseline
  Satisfaction questionnaire about the use of a telemedicine software

CONTACTS AND LOCATIONS:
Overall Officials: François Desmeules, Ph.D., Principal Investigator — CIUSSS Centre-Est-de-l"île-de-Montréal, Installation Maisonneuve-Rosemont Research Center
Locations (1):
- CIUSSS Centre-est-de-l'île-de-Montréal - Hopital Maisonneuve-Rosemont, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Doiron-Cadrin P, Kairy D, Vendittoli PA, Lowry V, Poitras S, Desmeules F. Feasibility and preliminary effects of a tele-prehabilitation program and an in-person prehablitation program compared to usual care for total hip or knee arthroplasty candidates: a pilot randomized controlled trial. Disabil Rehabil. 2020 Apr;42(7):989-998. doi: 10.1080/09638288.2018.1515992. Epub 2019 Jan 13. PMID 30638076
- [Derived] Doiron-Cadrin P, Kairy D, Vendittoli PA, Lowry V, Poitras S, Desmeules F. Effects of a tele-prehabilitation program or an in-person prehabilitation program in surgical candidates awaiting total hip or knee arthroplasty: Protocol of a pilot single blind randomized controlled trial. Contemp Clin Trials Commun. 2016 Oct 5;4:192-198. doi: 10.1016/j.conctc.2016.10.001. eCollection 2016 Dec 15. PMID 29736482